CLINICAL TRIAL: NCT01194206
Title: Downstaging of Hepatocellular Carcinoma by Stereotactic Body Radiotherapy for Non-Resectable and Non-Transplantable Tumors: Phase 2 Study
Brief Title: Stereotactic Body Radiation Therapy in Liver Cancer That Cannot be Removed by Surgery or Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study being rewritten
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3209; NCI-2010-01883 (Other: NCI/CTRP)
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo 3 fractions of stereotactic body radiation therapy in 3 fractions delivered within 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — At least 3 gold standard Cyberknife fiducials will be placed in the liver w/in 6 cm of the tumor for image guidance during radiation therapy. At least 1 wk will elapse between fiducial placement and tx planning simulation to allow for fiducial settling and any migration.The full radiation tx will be given ideally in 3 consecutive days. In any case there must be a minimum of 24 hrs between fractions and all 3 fractions will be delivered w/in 14 days. The dose to at least 95% of the tumor will be 37.5 Gy total in 12.5 Gy fractions.
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to kill tumor cells. Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue in patients with liver cancer. Giving stereotactic body radiation therapy may also increase patient eligibility for liver transplant.PURPOSE: This phase II trial is studying how well stereotactic body radiation therapy works in treating patients with liver cancer that cannot be removed by surgery or transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:I. To determine in patients with stage B and C Hepatocellular Carcinoma, if Stereotactic Body Radiotherapy can achieve a downstaging rate of >= 30% at 3 months.SECONDARY OBJECTIVES:I. To determine in patients with stage B and C Hepatocellular Carcinoma, if Stereotactic Body Radiotherapy can achieve a downstaging rate of >= 30% at 3 and 6 months.II. To determine the rate of Grade 3 or 4 adverse events associated with SBRT for liver tumors. III. To determine the rate of local progression after SBRT. (Based onRECIST criteria)IV. To determine the number of patients who achieve liver transplantation.OUTLINE:Patients undergo 3 fractions of stereotactic body radiation therapy delivered within 14 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* HCC is staged as Barcelona B or C (non-resectable and non-transplantable)
* Treatment with SBRT can occur within 6 weeks of staging laparoscopy
* Patient has a) Radiographic enhancing liver lesions on triple phase CT or MRI and b) Histological confirmation of HCC
* Patients with clinical/imaging features of HCC but without biopsy confirmation can be initially enrolled on the protocol and undergo staging laparoscopy for biopsy confirmation with the option of having the fiducials placed in the same procedure; but if the histology is not confirmed and/or other exclusion criteria is met patient will be taken off protocol
* Total aggregate of maximal dimension of liver tumors =< 8 cm
* Cirrhotic patients Child Pugh Class A or B
* Patient should be medically eligible for liver transplantation
* Absolute neutrophil count > 1,500/ul
* Platelets > 50,000 ul (after transfusion if required)
* Hemoglobin greater than 10.0 g/dL
* Total bilirubin < 2.0 mg/dL
* AST(SGOT)/ALT(SGPT) < 2 X institutional upper limit of normal
* Life expectancy > 12 weeks
* ECOG performance status < 2 or Karnofsky >= 70%
* Women of child-bearing potential must have a negative pregnancy test within 4 weeks to the start of the SBRT treatment
* Women must not be pregnant or nursing
* Sexually active men and women must agree to use accepted forms of birth control
* Provision of informed consent: Patient must be able to provide verbal and written informed consent

Exclusion Criteria:

* Patient with previous history of abdominal radiation
* Prior invasive malignancy other than primary liver malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Evidence of metastatic disease prior to staging laparoscopy
* Evidence of main Portal Vein thrombosis
* History of cardiac ischemia or stroke within last 6 months
* Any concurrent medical or psychosocial condition that prohibits a major surgical procedure or immunosuppression that would constitute a contraindication to liver transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Rate of downstaging of stage B and C Hepatocellular Carcinoma using Stereotactic Body Radiotherapy | At 3 months

SECONDARY OUTCOMES:
Rate of Grade 3 or 4 adverse events associated with SBRT for liver tumors as assessed by NCI CTCAE version 4.0 | Baseline, at 1 month, 3 months and 6 months
Rate of local progression as assessed by RECIST criteria | Baseline, at 1 month, 3 months and 6 months
Number of patients who achieve liver transplantation | at 6 months after SBRT
Survival rate | Survival will be measured from the first day of treatment on study until death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sanabria, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center